CLINICAL TRIAL: NCT07365956
Title: The Effect of Oral Care Using Apple Cider Vinegar, Chlorhexidine Gluconate and Sodium Bicarbonate on Oral Microbial Colonization in Neurosurgery Intensive Care Patients
Brief Title: Comparison of Oral Care Solutions on Oral Microbial Colonization in Neurosurgical ICU Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Harran University (Other)
Responsible Party: Principal Investigator, MURAT TAMER, Assistant Professor, Harran University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: HarranU-MTAMER-001
Record Dates: First submitted 2025-12-23; First posted 2026-01-26 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Oral Care
Keywords: Chlorhexidine Gluconate; Neurosurgery; Sodium Bicarbonate; nursing; apple cider vinegar
MeSH Terms: interventions — chlorhexidine gluconate; Sodium Bicarbonate

STUDY DESIGN:
Intervention Model Description: The patients in the experimental and control groups were determined using the Research Randomizer program (https://www.randomizer.org/). Before randomization, a drawing method was used to assign group numbers to the patients, designating 1 as the apple cider vinegar group, 2 as the chlorhexidine gluconate group, and 3 as the sodium bicarbonate group. Subsequently, numbers from 1 to 90 were randomized, and the groups were listed in order next to the numbers.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Chlorhexidine Gluconate Group (Experimental): Before Oral Care:
  The Patient Identification Form was filled out. The Oral Assessment Scale was applied. An oral culture sample was obtained.
  Procedure:
  Participants receive oral care using chlorhexidine gluconate solution every 6 hours for 5 days in the neurosurgical intensive care unit..
  The Oral Assessment Scale was applied. On the final day (Day 5), an oral culture sample was obtained.
  Interventions: Drug: Chlorhexidine gluconate (CHG)
- Sodium Bicarbonate Group (Experimental): Before Oral Care: The Patient Identification Form was filled out. The Oral Assessment Scale was applied. An oral culture sample was obtained. Procedure: Participants receive oral care using sodium bicarbonate solution every 6 hours for 5 days in the neurosurgical intensive care unit. The Oral Assessment Scale was applied. On the final day (Day 5), an oral culture sample was obtained.
  Interventions: Drug: Sodium Bicarbonate (NaHCO3)
- Apple Cider Vinegar Group (Experimental): Before Oral Care: The Patient Identification Form was filled out. The Oral Assessment Scale was applied. An oral culture sample was obtained. Procedure: Participants receive oral care using apple cider vinegar solution every 6 hours for 5 days in the neurosurgical intensive care unit. The Oral Assessment Scale was applied. On the final day (Day 5), an oral culture sample was obtained.
  Interventions: Other: Apple Cider Vinegar

INTERVENTIONS:
Drug: Chlorhexidine gluconate (CHG) — Oral care performed using chlorhexidine gluconate solution as part of routine oral hygiene in neurosurgical intensive care unit patients.
  Other Names: CHG
  Arms: Chlorhexidine Gluconate Group
Drug: Sodium Bicarbonate (NaHCO3) — Oral care performed using sodium bicarbonate solution to reduce oral microbial colonization in neurosurgical intensive care unit patients.
  Arms: Sodium Bicarbonate Group
Other: Apple Cider Vinegar — Oral care performed using diluted apple cider vinegar solution as an alternative oral hygiene intervention in neurosurgical intensive care unit patients.
  Arms: Apple Cider Vinegar Group

SUMMARY:
In the high-stakes environment of the Neurosurgery Intensive Care Unit (NSICU), patient stability extends beyond neurological monitors and intracranial pressure readings. A critical yet often underemphasized front line of defense is oral health. Neurosurgery patients, frequently intubated, on mechanical ventilation, or with depressed consciousness, are at extreme risk for Ventilator-Associated Pneumonia (VAP) and systemic infections. Pathogenic oral microbiota can be aspirated into the lower respiratory tract, triggering such complications. Consequently, rigorous oral care is not merely a comfort measure but a vital infection control protocol. This article examines and compares the effects of three agents-Chlorhexidine Gluconate (CHG), Sodium Bicarbonate, and Apple Cider Vinegar (ACV)-on oral microbial colonization in this vulnerable population.

DETAILED DESCRIPTION:
The normal oral flora undergoes a dramatic shift in critically ill patients. Factors like mouth breathing, nil-by-mouth status, decreased salivary flow, and the presence of endotracheal tubes create a pathogenic-friendly environment. This dysbiosis leads to colonization by opportunistic pathogens like Staphylococcus aureus, Pseudomonas aeruginosa, and Candida species. For neurosurgery patients, an ensuing pneumonia can lead to sepsis, increased intracranial pressure from systemic inflammation, prolonged ventilation, and longer ICU stays, directly impacting neurological recovery.

Aim of this study to examine the effect of oral care using ACV, chlorhexidine gluconate and sodium bicarbonate on oral microbial colonization in neurosurgery intensive care patients.

ELIGIBILITY:
Inclusion Criteria:

* Mechanical ventilation was initiated less than 24 hours ago,
* Aged 18 years or older,
* Had not undergone any oral surgical procedure,
* Were not leukopenic or thrombocytopenic,
* And had no oral infection such as aphthous ulcer, stomatitis, or gingivitis.

Exclusion Criteria:

* Mechanical ventilation was initiated more than 24 hours ago,
* Under 18 years of age,
* Had undergone any oral surgical procedure,
* Were leukopenic or thrombocytopenic,
* Or had an oral infection such as aphthous ulcer, stomatitis, or gingivitis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2022-01-01 (Actual); Study Completion 2022-01-01 (Actual)

PRIMARY OUTCOMES:
Change From Baseline in Oral Microbial Colonization Levels and Oral Assessment Scale Score | Day 0 to Day 5
  Oral microbial colonization will be measured using quantitative culture analysis of oral swab samples. Results will be reported as colony-forming units (CFU). The primary outcome is the change in CFU values from baseline (Day 0) to Day 5 following the oral care intervention.
  Oral mucosal condition will be measured using the Oral Assessment Scale. Scores will be recorded at baseline (Day 0) and on Day 5. The outcome will be reported as the change in total scale score between the two time points.
  All outcome measurements were completed within the first 5 days following initiation of the oral care intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Murat Tamer, Asst. Prof., Study Director — Harran University; Meral Ozkan, Professor, Principal Investigator — Inonu University
Locations (1):
- Inonu University, Malatya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No